CLINICAL TRIAL: NCT07379606
Title: A Comparison of Psychophysiological Effects Between Relaxation Techniques and Physical Exercise in Young Adults
Brief Title: Effects of Moderate Exercise and Cyclic Sighing on Stress, Cognition and Physiological Markers in Young Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 716/25
Record Dates: First submitted 2025-11-19; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Stress

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate-Intensity Physical Activity (PA) (Experimental): Participants perform 15 minutes of stationary cycling at moderate intensity.
  Interventions: Behavioral: Moderate-Intensity Physical Activity (PA)
- Breathing Training - Cyclic Sighing (CS) (Experimental): Participants perform 15 minutes of cyclic sighing.
  Interventions: Behavioral: Breathing Training - Cyclic Sighing (CS)

INTERVENTIONS:
Behavioral: Moderate-Intensity Physical Activity (PA) — Participants perform 15 minutes of stationary cycling at moderate intensity.
  Arms: Moderate-Intensity Physical Activity (PA)
Behavioral: Breathing Training - Cyclic Sighing (CS) — Participants perform 15 minutes of cyclic sighing (a breathing technique).
  Arms: Breathing Training - Cyclic Sighing (CS)

SUMMARY:
This study investigates the effects of moderate physical exercise and cyclic sighing (breathing training) on stress, cognition, and physiological markers in young adults. It is a randomized cross-over trial with two interventions. Each participant will take part in two intervention sessions:

1. Moderate-intensity physical activity (PA): 15 minutes of stationary cycling at 65-75% of maximum heart rate (HRmax).
2. Breathing training (CS): 15 minutes of cyclic sighing, a technique involving inhaling, pausing briefly, taking a deeper breath, and exhaling slowly.

A one-week washout period between sessions is planned to minimise carry-over effects and to ensure participants' physiological state is similar before the next session. During this week, participants will wear Polar Ignite wrist-worn devices to monitor physical activity and sleep.

A total of 30 participants (you adults) will be enrolled.

Measurements performed before and after each intervention include:

* EEG using Emotiv EPOC Flex Gel (32-channel device): 2 minutes with eyes open, 2 minutes with eyes closed, during the interventions, and while performing cognitive test (N-back).
* Heart rate variability (HRV) using the Polar H10 sensor.
* SUDS - Subjective Units of Disress Scale for perceived stress.
* N-back test for cognitive performance using Emotiv App.
* Blood pressure (systolic and diastolic) and heart rate.
* Pain threshold measured with a dolorimeter.
* PANAS-SF - Positive and Negative Affect Schedule.

Baseline questionnaires completed by participants the day before the study:

* PSS-10 - Perceived Stress Scale (Cohen, Kamarck, Mermelstein).
* MAAS - Mindful Attention Awareness Scale
* Psychological well-being - short version
* Mini-COPE - Coping with Stress Inventory
* Sleep quality and average sleep duration
* Chronotype questionnaire (morningness-eveningness)
* GPAQ - Global Physical Activity Questionnaire
* Pittsburgh Sleep Quality Index

The study aims to understand how brief interventions like moderate exercise and breathing techniques affect stress, cognitive performance, and physiological responses in young adults.

ELIGIBILITY:
Inclusion Criteria:

* male or female participants,
* age 18-35,
* without chronic somatic diseases,
* no current episode of psychiatric disorder (no active depression, mania, or psychosis),
* regular sleep schedule in the week prior to the study,
* not taking psychotropic drugs or medications,
* non-smoker,
* not working nightshifts.

Exclusion Criteria:

* consumption of alcohol or psychoactive substances the day before or on the day of the study,
* intense physical activity less than 2 hours before the study,
* consuming coffee, black tee, energy drinks less than 2 hours before the study,
* contraindications to moderate-intensity physical activity on cycle ergometer (e.g., recent injuries),
* contraindications to EEG (e.g., scalp skin conditions preventing proper electrode placement, hypersensitivity to conductive gels or pastes).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Mean EEG spectral power in theta, alpha, low beta, high beta, gamma frequency bands during resting-state (eyes-open and eyes-closed) | Baseline: immediately before intervention; Post-intervention: immediately after completion of the intervention period
  Mean spectral power in theta, alpha, low beta, high beta, and gamma frequency bands derived from resting-state EEG recordings collected during eyes-open and eyes-closed conditions. Spectral power will be calculated separately for eyes-open and eyes-closed resting-state conditions.
Heart Rate Variability (HRV) | Baseline (average over 5-minute resting-state immediately before intervention); During intervention (average over entire session, periprocedural); Post-intervention (average over 5-minute resting-state immediately after intervention).
  HRV will be recorded at three time points. Baseline HRV will be calculated as the average over a 5-minute resting-state period immediately before intervention. HRV during the intervention will be calculated as the average over the entire intervention session (periprocedural). Post-intervention HRV will be calculated as the average over a 5-minute resting-state period immediately after intervention.

SECONDARY OUTCOMES:
Mean EEG spectral power in theta, alpha, low beta, high beta, and gamma frequency bands during N-back task | Baseline (during N-back task immediately before each intervention session, periprocedural); Post-intervention (during N-back task immediately after each intervention session, periprocedural)
  Mean spectral power in theta, alpha, low beta, high beta, and gamma frequency bands derived from EEG recordings collected during performance of the N-back cognitive task. Spectral power will be calculated separately for each frequency band and averaged across all EEG channels.
Mean EEG spectral power in theta, alpha, low beta, high beta, and gamma frequency bands during intervention session | During intervention session (periprocedural, averaged over entire session)
  Mean spectral power in theta, alpha, low beta, high beta, and gamma frequency bands derived from EEG recordings collected during the intervention session. Spectral power will be calculated separately for each frequency band and averaged across all EEG channels.
Perceived Stress measured with the Subjective Units of Distress Scale (SUDS) | Baseline: immediately before each intervention session; Post-intervention: immediately after each intervention session
  Participants rate their perceived stress using the Subjective Units of Distress Scale (SUDS), a self-reported scale ranging from 0 (no stress) to 100 (extreme stress), where higher scores indicate higher perceived stress.
Cognitive Performance (N-back) | Baseline: immediately before each intervention session; Post-intervention: immediately after each intervention session
  Working memory assessed using N-back test with Emotiv app.
Blood Pressure | Baseline: immediately before each intervention session; Post-intervention: immediately after each intervention session
  Systolic and diastolic blood pressure measured using standard protocols.
Pain Threshold | Baseline: immediately before each intervention session; Post-intervention: immediately after each intervention session
  Pain threshold measured using a dolorimeter (algorimeter)
Positive and Negative Affect measured with the Positive and Negative Affect Schedule - Short Form (PANAS-SF) | Baseline: immediately before each intervention session; Post-intervention: immediately after each intervention session
  Participants complete the Positive and Negative Affect Schedule - Short Form (PANAS-SF), a self-reported scale assessing positive and negative affect. Each subscale contains 10 items rated from 1 (very slightly or not at all) to 5 (extremely), giving a possible score range of 10-50 for each subscale. Higher scores indicate higher levels of positive or negative affect, depending on the subscale.
Heart Rate | Baseline: immediately before each intervention session; Post-intervention: immediately after each intervention session
  Heart rate measured using standard protocols.

OTHER OUTCOMES:
Psychological Well-Being measured with the Short Version of Ryff's Psychological Well-Being Scale | Day before first intervention.
  Participants complete the Short Version of Ryff's Psychological Well-Being Scale, a self-reported questionnaire assessing psychological well-being across multiple dimensions. Items are rated on a scale from 1 (strongly disagree) to 6 (strongly agree), giving a total possible score range of 18-108, where higher scores indicate higher levels of psychological well-being.
Trait Mindfulness measured with the Mindful Attention Awareness Scale (MAAS) | Day before first intervention.
  Participants complete the Mindful Attention Awareness Scale (MAAS), a self-reported questionnaire measuring trait mindfulness. Items are rated on a scale from 1 (almost always) to 6 (almost never), with total scores ranging from 15 to 90. Higher scores indicate higher levels of trait mindfulness.
Coping with Stress measured with the Brief COPE Inventory (mini-COPE) | Day before first intervention.
  Participants complete the Brief COPE Inventory (mini-COPE), a self-reported questionnaire assessing coping strategies and stress management. Each item is rated on a scale from 1 (I haven't been doing this at all) to 4 (I've been doing this a lot), with total subscale scores ranging from 2 to 8, depending on the subscale. Higher scores indicate greater use of the specific coping strategy.
Chronotype measured with the Morningness-Eveningness Questionnaire (MEQ) | Day before first intervention.
  Participants complete the Morningness-Eveningness Questionnaire (MEQ) to assess chronotype, indicating morningness-eveningness preference. Items are scored to give a total score ranging from 16 to 86, where higher scores indicate greater morningness and lower scores indicate greater eveningness.
Global Physical Activity measured with the Global Physical Activity Questionnaire (GPAQ) | Day before first session.
  Participants complete the Global Physical Activity Questionnaire (GPAQ) to assess baseline physical activity levels. Responses are used to calculate total physical activity expressed in MET-minutes per week, with higher scores indicating higher levels of physical activity.
Sleep Quality and Duration (Pittsburgh Sleep Quality Index) | Day before first session.
  Participants complete the Pittsburgh Sleep Quality Index (PSQI) to assess sleep quality and average sleep duration.
Objective Sleep and Physical Activity (Polar Ignite) | During the 1-week washout period between intervention sessions.
  Participants wear Polar Ignite wrist-worn devices to monitor sleep quality and duration, as well as daily physical activity levels.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared in the RepOD repository after study completion. An embargo of up to 36 months may apply to allow for publication of primary study results. Data will be available for scientific research purposes.